CLINICAL TRIAL: NCT02540642
Title: Effect of Vitamin B12 Supplementation on Glycaemic Control in Uncontrolled Hyperhomocysteinemic Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smt. Kashibai Navale Medical College and General Hospital (Other)
Responsible Party: Principal Investigator, Dr Yogendra Keche, Associate Professor, Smt. Kashibai Navale Medical College and General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKNMC No./Ethics/App/2010/45
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes; Vitamin B12 Deficiency; Hyperhomocysteinemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin B 12 Deficiency; Hyperhomocysteinemia | interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin B12 and Antidiabetics (Active Comparator): Tablet Methylcobalamin 500 ug once daily with other usual antidiabetic drugs
  Interventions: Dietary Supplement: METHYLCOBALAMIN 500 micrograms
- antidiabetics (No Intervention): Only regular antidiabetic drugs will be given

INTERVENTIONS:
Dietary Supplement: METHYLCOBALAMIN 500 micrograms — Tab Methycobalamin 500 ug will be given with other regular antidiabetic drugs
  Other Names: Vitamin B12
  Arms: Vitamin B12 and Antidiabetics

SUMMARY:
Increased plasma homocysteine level is associated with macroangiopathy and nephropathy in type 2 diabetes. Also increased levels of serum homocysteine are associated with microalbuminuria which is associated with increased cardiovascular morbidity and mortality among the patients with type 2 diabetes. With B12 supplementation homocysteine level can be reduced .Type 2 diabetes as a metabolic syndrome may show improvement in glycaemic control with Vitamin B12 therapy as there is correction of hyperhomocysteinemia. In studies it is proved that combination of vit B12, folic acid and vit B6 are effective for hyperhomocysteinemia.There are no such separate trials on the use of vit B12 alone. This therapy may be used in large number of type 2 uncontrolled diabetic hyperhomocysteinemic patients.

this study was planned with following objectives to study effect of Vitamin B12 supplementation on glycaemic control in poorly controlled hyperhomocysteinemic type 2 diabetic patients

1. Glycaemic control measured by levels of glycosylated haemoglobin (HbA1c) at baseline and 4 weeks
2. Fasting blood sugar level at baseline and 4 weeks
3. Serum homocysteine/ vitamin B12 levels at baseline and 4 weeks
4. Serum lipid profile at baseline and 4 weeks

DETAILED DESCRIPTION:
After approval from Institutional Ethics Committee, patients not responding adequately to oral anti-diabetic agents were recruited from Medicine out patient department (OPD) with the help of treating physician. Patient were first screened for serum homocysteine/vitamin B12 level along with all baseline investigations. Those having serum homocysteine level more than 15 umol/L or vitamin B12 level less than 223pg/ml were enrolled in this study. Due to high cost for investigation serum homocysteine level was measured only in 6 patients and serum vitamin B12 level (cheaper test) was measured in 14 patients with prior permission from Ethics Committee. Patients were given all the information about Vitamin B12 (methylcobalamin) including adverse effects. A written informed consent was taken from each patient and those who were willing to participate in study were enrolled in this study. All the information was recorded in case report forms.

There were two groups of poorly controlled patient; one group (DRUG GROUP) received methylcobalamin 500 ug daily with their usual antidiabetic therapy and the other group (CONTROL GROUP) received suitable antidiabetic drug therapy as prescribed by treating physician. Methylcobalamin 500ug was given once daily for the period of 4 weeks and were followed-up at 4 weeks. At Baseline all the investigations were carried out as follows:

Study Flow Chart

Baseline Serum Homocysteine.n=6 (DRUG GROUP), Serum Vitamin B12, n=14 (DRUG GROUP), n=18 (CONTROL GROUP) Body weight, height, Blood pressure,glycosylated hemoglobin (HbA1c) level, Blood sugar-Fasting/Postprandial, Serum lipid profile( to measure the effect of Vitamin B12), Blood urea, Serum creatinine, Serum Bilirubin, Serum glutamate oxaloacetate transaminase (SGOT),Serum glutamate pyruvate transaminase (SGPT), Alkaline phosphatase ( to rule out hepatic or renal dysfunction ), Routine urine examination for albumin, Electrocardiogram (ECG):to rule out cardiac abnormality viz, IHD, arrhythmias

4 Weeks Body weight, Blood pressure, glycosylated hemoglobin(HbA1c) level, Blood sugar-Fasting/Postprandial, Serum lipid profile, Serum homocysteine/ serum vitamin B12, Urine albumin examination

After enrollment of patient for study, All the baseline investigations will be carried out at Central Clinical Laboratory except glycosylated haemoglobin which was carried out at department of Pharmacology and homocysteine estimation which was carried out in an accredited laboratory. ECG, Blood pressure recording was carried out in Department of Medicine.

Reporting of Adverse effects: All patients had been given checklist of adverse effect of vitamin B12. Information of adverse drug reactions (ADRs ) was taken in next follow-up. If patients are unable tolerate adverse drug reactions they were advised to contact any of investigators at any time. Contact numbers of investigators was mentioned on patient information sheet.

Expected adverse drug reactions of vitamin B12 : Anorexia, Nausea, Vomiting, Diarrhea and Rash

Sample Size Calculation and statistical analysis:

Sample size of 20 for each group was calculated in the ratio of 1, power 80 %, considering 10 fold difference of drug effect in vitamin B12 group and control group by using Open Epi 2.3(2009). Randomization was done with the help of randomization software Rando 1.2,2004. Statistical analysis was done by using Open Epi 2.3(2009) and Microsoft Excel.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30 -70 years
2. Sex: Male/ Non-lactating female
3. Glycosylated hemoglobin (HbA1c) > 8
4. Serum Homocysteine > 15 umol / L or vitamin B12 less than 223pg/ml

Exclusion Criteria:

1. Age < 30 yrs.
2. Pregnancy
3. Lactating mother
4. Patient with Insulin dependent diabetes mellitus
5. Severe and Complicated diabetes mellitus
6. Patient with hepatic or renal dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To compare the change in HbA1c levels (%) with vitamin B12 supplementation in poorly controlled type 2 diabetic patients | baseline and 4 weeks

SECONDARY OUTCOMES:
To compare the change in high density lipoprotein(HDL),low density lipoprotein(LDL) and total cholesterol in mg/dL with vitamin B12 supplementation in poorly controlled type 2 diabetic patients | baseline and 4 weeks
To compare the change in fasting and postprandial blood sugar levels (mg/dL) with vitamin B12 supplementation in poorly controlled type 2 diabetic patients | baseline and 4 weeks
To compare the change in serum homocysteine level (micromol/L) with vitamin B12 supplementation in poorly controlled type 2 diabetic patients | baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: YOGENDRA N KECHE, MD, Principal Investigator — SMT KASHIBAI NAVALE MEDICAL COLLEGE
Locations (1):
- Smt Kashibai Navale Medical College and Hospital, Pune, Maharashtra, India